CLINICAL TRIAL: NCT02876744
Title: Correlation Between Macular Ischemia and Peripheral Ischemia in Patients With Diabetes
Acronym: CORISMAP
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: MMT_2016_21
Record Dates: First submitted 2016-08-19; First posted 2016-08-24 (Estimated); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: ophthalmologic examination — ophthalmologic examination including optical coherent tomography with angiography module

SUMMARY:
The contribution of OCT- angiography (OCT-A) allows to consider, in a more or less long term, a drastic reduction in the use of fluorescein angiographies in diabetic retinopathy. The accuracy of the analysis of the vascularization of retinal layers of the posterior pole of the eye by the OCT-A , will detect, early and in a quantifiable manner, whether or not there are areas of macular ischemia in a patient. However, current technical limitations (small field analysis) of OCT-A imaging only allow a limited study of retina at the posterior pole of the fundus.

This study seeks to demonstrate whether there is a link between macular ischemia detected by the OCT-A and peripheral retinal ischemia detected by the fluorescein angiographies, in diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* diabetes type I or type II
* follow-up with fluorescein angiography

Exclusion Criteria:

* known allergy to fluorescein
* contra-indication to fluorescein angiography
* pregnant or breast-feeding patient
* technical impossibility to analyse retinal ischemic areas on fluorescein angiography or OCT-A.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diabetes, requiring follow-up with fluorescein angiography.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2020-04-13 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Detection and measure of ischemic territories in central and peripheral retina | immediate

CONTACTS AND LOCATIONS:
Overall Officials: Martine MAUGET FAYSSE, MD, Principal Investigator — Fondation ophtalmologique de Rothschild
Locations (1):
- Fondation Opthalmologique A de Rothschild, Paris, France

IPD SHARING:
Plan to Share IPD: No